CLINICAL TRIAL: NCT02718196
Title: Testing and Development of a Sleep Training Mobile Health Application to Address Sleep Problems in the First Two Years of Life
Brief Title: Testing and Development of a Sleep Training Mobile Health Application
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: App stopped development before minimum viable product created
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1603017350
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application Users (Experimental): English-speaking parents of children ages 6-24 months who are interested in starting sleep training within the next month.
  Interventions: Behavioral: Sleep Training smartphone application

INTERVENTIONS:
Behavioral: Sleep Training smartphone application — Every evening the application provides a list of the planned bedtime activities as well as the recommended bedtime. The steps are 1) positive bedtime routine 2) bedtime fading 3)addressing nocturnal feeding 4) extinction protocol

SUMMARY:
The specific aims of this study are : 1) To pilot test the alpha build prototype of the sleep training smartphone application using a sample of parents looking for sleep training advice online. 1a) To assess the efficacy of the application in helping parents with the sleep training process 1b) To assess the 'workability' of the application 2) Use feedback to guide the next round of development with the goal of building out the applications functionality and increasing usability.

DETAILED DESCRIPTION:
Problems with bedtime and night-wakings are common in early childhood. Behavioral interventions to address these sleep problems are commonly referred to as "sleep training" and are effective but difficult for some parents to perform. The investigators have developed a prototype of a novel smartphone application designed to assist parents throughout this process.

The smartphone application first collects basic information from the parents, including: first name of child, number of caregivers participating in bedtime, tolerance of caregivers for crying, and basic information about timing of sleep and wake, as well as information about the usual order of events at bedtime. At each step, a brief (2-3 paragraph) is provided to explain the rationale for the next step, as well as concrete advice on how to succeed. It then walks parents through proven techniques to improve sleep in children in a stepwise fashion.

ELIGIBILITY:
Inclusion Criteria:

* english speaking
* parent of child age 6-24 months
* target child sleeping in crib in his or her own room (not the same room as the parents or a sibling)
* actively looking to sleep train their child
* own an iOS or Android smartphone

Exclusion Criteria:

* bedsharing/cosleeping with child
* target child has a known developmental delay
* target child has a significant health issue affecting his/her sleep (failure to thrive, congenital heart disease, etc).

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in average number of night wakings by Brief Infant Sleep Questionnaire (BISQ) | study entry and 1 month
  The question is: Average number of night wakings per night: ____________
  Brief Infant Sleep Questionnaire (BISQ)This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency.
Change in average number of night wakings by Brief Infant Sleep Questionnaire (BISQ) | study entry and 3 months
  Brief Infant Sleep Questionnaire (BISQ)This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Average number of night wakings per night: ____________
Perception of child's sleep problem- Brief Infant Sleep Questionnaire (BISQ) | study entry
  Brief Infant Sleep Questionnaire (BISQ)This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Do you consider your child's sleep as a problem?
  □ A very serious problem □ A small problem □ Not a problem at all
Perception of child's sleep problem- Brief Infant Sleep Questionnaire (BISQ) | 3 months
  Brief Infant Sleep Questionnaire (BISQ)This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Do you consider your child's sleep as a problem?

IPD SHARING:
Plan to Share IPD: No